CLINICAL TRIAL: NCT05130892
Title: Effect of Inflammasome Inhibitor on High-sensitivity C-reactive Protein in Patients After Percutaneous Coronary Intervention
Brief Title: Effect of Inflammasome Inhibitor on hsCRP in Patients After PCI
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Union Hospital, Tongji Medical College, Huazhong University of Science and Technology (Other)
Responsible Party: Principal Investigator, Xiang Cheng, Director of Cardiology, Union Hospital, Tongji Medical College, Huazhong University of Science and Technology, Union Hospital, Tongji Medical College, Huazhong University of Science and Technology
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: NLRP3-CRP
Record Dates: First submitted 2021-11-20; First posted 2021-11-23 (Actual); Last update posted 2023-02-08 (Actual); Status verified 2023-02

CONDITIONS: NLRP3; hsCRP; Percutaneous Coronary Intervention
MeSH Terms: interventions — Colchicine; tranilast; oridonin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Colchicine group (Experimental): 1 tablet (0.5mg) / time, once a day
  Interventions: Drug: Colchicine
- Tranilast group (Experimental): 1 capsule (0.1g) / time, 3 times a day;
  Interventions: Drug: Tranilast
- Oridonin group (Experimental): 2 tablets (0.5g) / time, 3 times a day
  Interventions: Drug: Oridonin
- Non-intervention group (No Intervention)

INTERVENTIONS:
Drug: Colchicine — 1 tablet (0.5mg) / time, once a day
  Arms: Colchicine group
Drug: Tranilast — 1 capsule (0.1g) / time, 3 times a day
  Arms: Tranilast group
Drug: Oridonin — 2 tablets (0.5g) / time, 3 times a day;
  Arms: Oridonin group

SUMMARY:
Coronary artery disease (CAD) comprises the major contributor to a global epidemic of cardiovascular disease. Patients with CAD undergoing percutaneous coronary intervention (PCI) have a high-risk for adverse clinical outcomes.

Residual inflammatory risk (RIR) in patients with CAD after standardized treatment is the main cause of adverse events such as recurrent myocardial infarction, stroke, and death, which has gained much interest in recent years. Inflammation plays an important role in the development of CAD. However, several randomized controlled clinical studies (RCT) of anti-inflammatory treatments ended in failure previously. Since 2017, the success of three large-scale RCTs (CANTOS, COLCOT and LoDoCo2) points to targeting the NLRP3 - IL-1 β- IL-6 pathway for anti-inflammatory treatment of CAD. The inhibition of this pathway eventually leads to the decrease of high-sensitivity C-reactive protein (hsCRP), consistent with an anti-inflammatory effect. Therefore, the change of hsCRP may serve as a biomarker to screen anti-inflammatory drugs in this pathway.

Targeting the NLRP3 - IL-1 β- IL-6 pathway with monoclonal antibodies is limited by high prices of the biological agents. Thus, researchers focused on the upstream molecule NLRP3. Currently, NLRP3 inhibitors that are clinically available include colchicine , tranilast and oridonin. Although several studies have indicated the effective effects of colchicine in CAD, the other two NLRP3 inhibitors lack sufficient data on anti-inflammatory treatment of CAD. Therefore, we intend to use NLRP3 inhibitors (colchicine, tranilast and oridonin) to treat patients after PCI for 4 weeks, compare the changes of hsCRP, and explore the effectiveness and safety of these different drugs, and screen the optimal anti-inflammatory drugs for coronary heart disease.

ELIGIBILITY:
Inclusion Criteria:

1. Voluntarily participate, and sign the informed consent form;
2. Age ≥ 18 and ≤ 80 years, regardless of sex;
3. Patients after completion of planned percutaneous coronary intervention for 4 weeks.

Exclusion Criteria:

1. Allergic to colchicine, tranilast or oridonin;
2. Taking colchicine, tranilast or oridonin before the screening period (10 days);
3. Abnormal liver function (ALT > 3 times the upper limit of normal value);
4. Abnormal renal function (creatinine clearance < 45 ml / min);
5. Thrombocytopenia (PLT < 100g / L);
6. Uncontrolled infectious diseases;
7. Complicated with immune diseases or immune related diseases such as systemic lupus erythematosus, asthma, inflammatory bowel disease, gout, and malignant tumor, etc.
8. Nonsteroidal anti-inflammatory drugs, hormones, immunomodulatory and chemotherapeutic drugs been taken;
9. History of surgery within 6 months before the screening period;
10. Pregnant women, lactating women or women of childbearing age who do not use effective contraceptives;
11. Other circumstances in which the investigator judges that the patient is not suitable to participate in the clinical trial.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 132 (Actual)
Dates: Start 2021-11-15 (Actual); Primary Completion 2023-02-01 (Actual); Study Completion 2023-02-01 (Actual)

PRIMARY OUTCOMES:
Percentage change in hsCRP | 4 weeks
  Percentage change in hsCRP at the end of 4 weeks compared with baseline

SECONDARY OUTCOMES:
MACE (composite endpoint of all-cause death, nonfatal myocardial infarction, nonfatal stroke, revascularization due to ischemia, or hospitalization due to unstable angina pectoris) | 4 weeks
  Time to occurrence of MACE
Bleeding | 4 weeks
  Time to occurrence of bleeding
Proteomics analysis | 4 weeks
  Proteomics analysis using cardiovascular II/III panel by Olink company

CONTACTS AND LOCATIONS:
Locations (2):
- China (2):
  - Department of Cardiology, Union Hospital, Tongji Medical College, Huazhong University of Science and Technology, Wuhan, Hubei
  - Wuhan Union Hospital, Wuhan, Hubei

IPD SHARING:
Plan to Share IPD: No